CLINICAL TRIAL: NCT06207149
Title: Adapting an Advocacy Services Intervention for Latinx Families of Transition-aged Youth With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Meghan Burke, Professor, Special Education, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R03MH129757-01A1 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2024-01-16 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will attend an advocacy program.
  Interventions: Behavioral: ASISTIR
- Waitlist-Control Group (Active Comparator): Participants will receive the written materials of the advocacy program. After completing the intervention group completes the advocacy program, the waitlist-control group participants will be able to participate in the advocacy program.
  Interventions: Behavioral: ASISTIR

INTERVENTIONS:
Behavioral: ASISTIR — This will be a 24 hour advocacy program focused on adult disability services.

SUMMARY:
When youth with autism spectrum disorder (ASD) transition from school to adult services, they fall off a "service cliff." To increase access to services, the investigators developed the ASSIST program, which teaches parents how to advocate for adult services on behalf of youth with ASD. In a pilot randomized controlled trial (RCT: R34 MH104428), treatment group (versus control) participants demonstrated significantly improved knowledge of adult services, advocacy, and empowerment. Sons/daughters of treatment group participants had increased access to services. For advocacy services interventions like ASSIST to be equitable, they need to reach families who are at greatest risk for service disparities. Latinx youth with ASD are one such underserved population. Relative to White youth, Latinx youth with ASD receive significantly fewer post-secondary education, health, and employment services and face worse post-school outcomes. In addition to the barriers which hinder service access for all families, Latinx families face unique barriers to service access (e.g., language, cultural differences, citizenship, discrimination) making them a marginalized population. In this project, the investigators are adapting the ASSIST curriculum and related measures for Latinx parents of transition-aged youth with ASD. Specifically, the investigators will leverage ASSIST data and data from Latinx, non-ASSIST parents to inform adaptations to the ASSIST curriculum. The investigators will also conduct pre-testing and a cross-cultural adaptation process to revise the ASSIST measures for Latinx families. The investigators will test the adapted ASSIST curriculum with a randomized controlled trial to determine its feasibility, acceptability and efficacy on intervention targets (knowledge, advocacy, and empowerment) and outcome of interest (service access). This project is aligned with NIMH priorities by examining services from adolescence to adulthood (PA-21-199) and by adapting a program to improve mental health services for underserved populations NIMH 2020 Strategic plan). It is also responsive to the Interagency Autism Coordinating Committee core value of "equity" in reducing disparities with respect to cultural backgrounds. Further, if successful, it will be the first intervention to directly address service disparities for Latinx families of youth with ASD who are transitioning to adulthood.

ELIGIBILITY:
Inclusion Criteria: To be included in the study, the participant must be:

* over the age of 18,
* identify as Latinx,
* have a child with autism who is over the age of 12,
* speak Spanish, and
* reside in Illinois.

Exclusion Criteria:

* Must understand Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to upload de-identified data to NDAR.

REFERENCES:
- [Derived] Burke MM, Ramos-Torres S, Espinosa GH, Hincapie AL, Aleman-Tovar J, Perez R, Puente C. Testing an Advocacy Program to Improve Service Access Among Latino Families of Autistic Youth: A Randomized Controlled Trial. Autism Res. 2025 Aug;18(8):1714-1724. doi: 10.1002/aur.70068. Epub 2025 Jun 21. PMID 40542546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Waitlist-Control Group
Started | 24 | 24
Completed | 17 | 13
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Waitlist-Control Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.75 (9.35) | 44.72 (6.12) | 44.74 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 48
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
Adult Disability Services Knowledge [Mean (Standard Deviation); unit: units on a scale] — A multiple-choice, multi-item scale assessing knowledge about adult disability services. Higher scores indicate greater knowledge (thus, higher scores are considered better outcomes). The scale ranges from 0 (minimum) to 24 (maximum). Unabbreviated scale title is Knowledge. The construct it measures is knowledge of adult disability services.
  units on a scale | 5.71 (4.35) | 4.16 (3.27) | 4.94 (4.09)
Individual Advocacy Activities [Mean (Standard Deviation); unit: units on a scale] | 18.50 (6.05) | 16.21 (3.55) | 16.43 (5.01)
Advocacy Skills and Comfort [Mean (Standard Deviation); unit: units on a scale] | 26.72 (8.35) | 28.21 (6.40) | 28.04 (8.500)
Family Empowerment [Mean (Standard Deviation); unit: units on a scale] | 47.27 (7.69) | 44.21 (7.15) | 46.43 (7.75)
Services Empowerment [Mean (Standard Deviation); unit: units on a scale] | 46.54 (8.84) | 43.89 (7.78) | 45.59 (8.46)
Community Political Empowerment [Mean (Standard Deviation); unit: units on a scale] | 30.72 (7.25) | 29.94 (6.78) | 30.29 (6.34)
Number of Services Received [Mean (Standard Deviation); unit: units on of measure of services] | .55 (.88) | 1.00 (1.19) | .67 (1.0)
Unmet Service Needs [Mean (Standard Deviation); unit: units on a scale] | 1.33 (2.24) | 1.63 (1.69) | 1.61 (2.23)

OUTCOME MEASURES:

1. Primary Outcome: Disability Knowledge Scale
Description: A multiple-choice, multi-item scale assessing knowledge about adult disability services. Higher scores indicate greater knowledge (thus, higher scores are considered better outcomes). The scale ranges from 0 (minimum) to 24 (maximum). Unabbreviated scale title is Knowledge. The construct it measures is knowledge of adult disability services.
Time Frame: Pre, Post (three months after the Intervention group takes the training), and Follow-up (six months after the intervention group takes the training).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist-Control Group
Number analyzed (Participants) | 17 | 13
units on a scale
  Post Survey | 10.62 (2.57) | 3.68 (4.59)
  Follow-up Survey | 6.84 (4.23) | 3.04 (3.45)

2. Primary Outcome: Advocacy Activities Scale
Description: A scale with three subscales assessing individual, peer, and systemic advocacy. Only individual advocacy was expected to increase. Higher scores indicate greater advocacy (thus, higher scores means better outcomes). The scale ranges from 12 (minimum) to 60 (maximum). Unabbreviated scale title is Advocacy. The construct the scale measures is advocacy.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist-Control Group
Number analyzed (Participants) | 17 | 13
units on a scale
  Post Survey | 20.00 (5.77) | 15.61 (5.28)
  Follow Up Survey | 33.75 (7.49) | 16.69 (4.63)

3. Primary Outcome: Family Empowerment Scale-Family Subscale
Description: The Family Empowerment Scale (the full scale name) measures the constructs of empowerment in relation to the family, community, and service delivery system.Higher scores indicate greater empowerment (thus, higher scores means a better outcome). The scale ranges from 12 (minimum) to 60 (maximum). The items are summed to create a total score. Unabbreviated scale title is Family Empowerment. The construct that the Family Subscale measures is empowerment within the family.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist-Control Group
Number analyzed (Participants) | 17 | 13
units on a scale
  Post Survey | 47.27 (7.69) | 44.21 (7.15)
  Follow-up Survey | 51.38 (8.36) | 46.62 (9.38)

4. Primary Outcome: Unmet Service Scale
Description: A scale measuring the extent of service needs among individuals with autism. Scores range from 0 (minimum)-16 (maximum) with higher scores indicating more unmet service needs (thus, lower scores are better outcomes). Unabbreviated scale title is Unmet Services. The construct is unmet service needs.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist-Control Group
Number analyzed (Participants) | 10 | 13
units on a scale
  Post survey | 1.00 (3.00) | .75 (1.49)
  Follow up Survey | 1.89 (1.96) | 3.12 (1.80)

5. Primary Outcome: Family Empowerment Scale-Service Delivery System Subscale
Description: The Family Empowerment Scale (the full scale name) measures the construct of empowerment in relation to the family, community, and service delivery system.Higher scores indicate greater empowerment (thus, higher scores means a better outcome). The scale ranges from 12 (minimum) to 55 (maximum). The items are summed to create a total score. Unabbreviated scale title is Services Empowerment. The construct this subscale measures is empowerment within the service delivery system.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist-Control Group
Number analyzed (Participants) | 17 | 13
units on a scale
  Post Survey | 47.31 (5.89) | 42.32 (11.16)
  Follow-up Survey | 51.00 (8.73) | 46.61 (9.38)

6. Primary Outcome: Family Empowerment Scale-Community and Political Subscale
Description: The Family Empowerment Scale (the full scale name) measures the constructs of empowerment in relation to the family, community, and service delivery system.Higher scores indicate greater empowerment (thus, higher scores means a better outcome). The scale ranges from 12 (minimum) to 55 (maximum). The items are summed to create a total score. Unabbreviated scale title is Community and Political Empowerment. The construct that the Community and Political Subscale measures is empowerment within the community and political contexts.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist-Control Group
Number analyzed (Participants) | 17 | 13
units on a scale
  Post Survey | 37.23 (7.13) | 29.62 (8.45)
  Follow-up Survey | 37.50 (7.25) | 33.31 (5.83)

7. Primary Outcome: Advocacy Skills and Comfort
Description: The full name of this measure is Advocacy Skills and comfort. The Advocacy Skills and comfort scale measures the construct of comfort with advocacy skills. The scale ranges from 10 to 50. Higher scores are better indicating greater comfort with advocacy skills. The items are summed to create a composite.
Time Frame: as for outcome 1
Population: Participants were compared by group assignment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention | Waitlist-Control Group
Number analyzed (Participants) | 17 | 13
Units on a scale
  Post Survey | 33.92 (8.42) | 25.38 (9.51)
  Follow-up | 33.75 (7.49) | 29.23 (9.01)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the study which was 24 months.
Description: There were no adverse events.
Arm/Group | Intervention | Waitlist-Control Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT06207149/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT06207149/SAP_001.pdf